CLINICAL TRIAL: NCT00733356
Title: The Effects of Vyvanse(TM) on Brain Hemodynamics and Reading
Acronym: VBHR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kimberley Lakes (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor-Investigator, Kimberley Lakes, Associate Professor, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: VBHR
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; ADD; reading; brain hemodynamics; brain imaging; attention; Near-Infrared Spectroscopy; NIRS; MSIT
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vyvanse Treatment (Experimental): All subjects were tested at baseline before medication and then titrated to best dose and retested on Vyvanse Medication.
  Interventions: Drug: Vyvanse

INTERVENTIONS:
Drug: Vyvanse — Subjects will participate in an open-label dose optimization period and successful titration to an optimal dose of Vyvanse™, subjects will take their optimized dose of Vyvanse™ (30, 50 or 70 mg/day) during the week leading up to their final visit. During the study subjects will take their prescribed dose once a day in the morning with breakfast.
  Other Names: lisdexamfetamine dimesylate

SUMMARY:
This is a single-blind, Investigator Initiated study to evaluate the safety and efficacy of Vyvanse™ and provide pilot data in two areas: (1) on the use of Near-Infrared Spectroscopy to detect medication effects in children with ADHD; and (2) on the influence of Vyvanse ™ on reading fluency and comprehension, over a period of approximately 6-8 weeks. Subjects will be between the ages of 6 and 12 at the beginning of the study.

DETAILED DESCRIPTION:
This is a single-blind study to evaluate the safety and efficacy of Vyvanse™ and provide pilot data in two areas: (1) on the use of Near-Infrared Spectroscopy to detect medication effects in children with ADHD; and (2) on the influence of Vyvanse ™ on reading fluency and comprehension over a period of approximately 6 weeks. Subjects will be between the ages of 6 and 12 at the beginning of the study.

The study will consist of periods detailed below:

Screening and Washout. Subjects will be screened up to four weeks prior to baseline. The washout period will be 3 days for most ADHD stimulant medication (the half life is around 3-5 hours and the washout is at least 5 half-lives in duration). Other medication will be discussed during the visit.

The Screening Visit will occur at the UCI Child Development Center and will allow for the determination of appropriateness of each subject's inclusion into the study. The Principal Investigator or his/her designee must obtain written signed and dated consent for the subject to participate in the study from the subject's parent(s)/legally authorized representative and assent must be given by the subject, prior to any study related procedures being performed. This visit is expected to last 3-4 hours and may take place across more than one day.

The following procedures will be conducted during the Screening Visit:

* Informed Consent/Assent obtained
* Psychiatric evaluation that utilizes the Kiddie-Schedule for Affective Disorders and Schizophrenia-Present and Lifetime Version (K-SADS-PL) and according to DSM-IV-TR™ criteria
* Inclusion/Exclusion criteria confirmed
* Demographics collected
* Medical and Medication History
* Physical Examination including height (using a calibrated stadiometer), weight (using a calibrated scale)
* Sitting Vital Signs after 5 minutes of rest (oral or tympanic temperature, pulse, blood pressure, and respiratory rate)
* 12-Lead ECG after 5 minutes of rest
* Kaufman Brief Intelligence Test 2 (KBIT2): used to assess both verbal and non-verbal cognitive ability.
* Concomitant Medications reviewed
* Adverse Events reviewed

In addition, the subject will be asked to give a small blood sample, for safety screening purposes, for laboratory procedures (approximately 2 teaspoons).The following lab procedures will be performed:

* Hematology with complete blood count (CBC)
* Serum Chemistry
* Urinalysis and microscopic examination (if protein and/or blood are detected during urinalysis)
* Serum Pregnancy Test for all FOCP - A negative serum pregnancy test must be documented for inclusion into this study
* Urine drug test Baseline Procedures. After all Screening and washout procedures have been completed, subjects will return to the site for the Baseline Visit, which will last approximately 5-6 hours.

Subjects will be provided with a one-week supply of VyvanseTM 30mg/day. Subjects will begin treatment the morning of the baseline visit and continue on the same dose for the next week. The first dose of medication will be administered on site and subsequent dosing will be given to the subject's parent(s)/legally authorized representative who will be required to administer study drug to the subject upon awakening. During the visit subjects will perform the Attention Task while the NIRS is recording and they will also be given the Gray's Oral Reading Test before the medication is administered. After the medication is administered the subject will stay on site until the second NIRS measurement can be taken a second time. They will be provided food and activities during the waiting period.

The following procedures will be conducted during the Baseline Visit:

* Confirmation of continued eligibility (i.e., with respect to inclusion/exclusion criteria and medication history)
* Sitting Vital Signs (oral or tympanic temperature, pulse, blood pressure and respiratory rate)
* Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent: Investigator Administered and Scored (ADHDRS-IV-Parent:Inv): The primary efficacy measure, used to assess the 18 symptoms of ADHD.
* Clinical Global Impressions Severity scale (CGI-S): This measure is used to assess the severity of the subject's symptoms.
* Concomitant Medications will be reviewed with the subject.
* Adverse Events
* Medication administered on-site
* Near Infrared Spectroscopy and Attention Task performed twice, once at before medication and again 3-4 hours after first exposure to medication.
* Administer the Gray Oral Reading Test-4 (GORT-4), which used to test oral reading rate, accuracy, fluency, and comprehension, before exposure to medication.
* Distribute Open-Label Study Drug - A one-week supply of VyvanseTM 30mg capsules will be dispensed, including the dose administered on site.

Dose Optimization. During the dose optimization period, subjects will visit the office once per week so that the study doctor can determine if the subject is tolerating the study medication and if she/he is seeing any benefit. These visits will last approximately 45 minutes. The Investigator will review AEs, ADHD-RS-IV, and CGI-I scores, and use clinical judgment to ensure that subjects are titrated to an acceptable dose of VyvanseTM for evaluation.

The following procedures will be conducted at each dose optimization visit:

* Sitting Vital Signs (oral or tympanic temperature, pulse, blood pressure and respiratory rate)
* Subject Weight (using a calibrated scale)
* Investigator Dose Assessment
* ADHD-RS-IV
* Clinical Global Impressions Improvement Scale (CGI-I).
* Study Drug Accountability and Compliance Assessment Performed
* Distribute Open-Label Study Drug
* Concomitant Medications
* Adverse Events Dose Optimized NIRS and GORT Testing

This visit will be similar to the baseline visit. Subjects will arrive early in the morning and medication will be administered on-site. They will remain on site for the next 4 hours so that the dose will be at peak effect before administering the GORT or NIRS. The following procedures will happen during this visit:

* Sitting Vital Signs after 5 minutes of rest (oral and tympanic temperature, pulse, blood pressure and respiratory rate)
* Subject weight (using a calibrated scale)
* An electrocardiogram will be performed.
* Serum Pregnancy Test for all FOCP - A negative serum pregnancy test must be documented for the end of the study.
* ADHD-RS-IV
* CGI-I
* Study Drug Accountability and Compliance Assessment Performed
* Concomitant Medications
* Adverse Events
* Medication administered on-site
* Near Infrared Spectroscopy and Attention Task performed once.
* Administer the Gray's Oral Reading Test.
* Physical examination including height (using a calibrated stadiometer)
* 12 Lead ECG 30-day Follow-up Phone Call

ELIGIBILITY:
Inclusion Criteria:

1. Females of child-bearing potential must have a negative pregnancy test.
2. Subjects must meet DSM-IV-TR™ criteria for a primary diagnosis of ADHD.
3. Subjects must have an ADHDRS-IV-Parent: Inv total score at least 1.5 standard deviations above the age and gender norms.
4. The subject is functioning at an age appropriate level intellectually as determined by an IQ score of ≥ 80 on the Kaufman Brief Intelligence Test.
5. The subject and subject's parent or legal guardian must be willing and able to comply with all the testing and dosing requirements in this study.
6. Subject has blood pressure measurements within the 95th percentile for age, gender, and height.
7. All subjects and their parents must be able to communicate effectively in English with the doctor and his/her staff without the aid of an interpreter.

Exclusion Criteria:

1. Subject has any documented, current, controlled psychiatric illness [except Oppositional Defiant Disorder (ODD)]. The child may continue participating in a behavior modification program during this study as long as he/she has been participating in the program for at least one month at the time of the baseline visit.
2. Subject has Conduct Disorder (CD).
3. Subject has a documented allergy, hypersensitivity or intolerance to amphetamines, which is the class of drug to which Vyvanse™ belongs.
4. Subject has failed to respond to one or more adequate courses (dose and duration) of amphetamine therapy.
5. Subject has a recent history (within the past 6 months) of suspected substance abuse or dependence disorder (excluding nicotine).
6. Subject had a history of seizures during the last two years (exclusive of febrile seizures), a tic disorder, or a current diagnosis and/or family history of Tourette's Disorder.
7. Subject has a history of heart abnormalities that the study doctor feels would exclude him/her from the study.
8. Subject has a positive urine drug result at the screening visit.
9. Subject weighs less than 50 pounds (22.7 kg).
10. Subject has taken another investigational drug within the last 30 days prior to the screening visit.
11. Subject has any reported history of abnormal thyroid function.
12. Subject has any clinically significant electrocardiogram reading (an electrical recording of the heart - ECG) or laboratory abnormalities at the screening and/or baseline visits.
13. The study doctor feels that the subject's safety would be jeopardized if entered in this study due to a current illness or medical condition. Mild, stable asthma is not exclusionary.
14. Subject is taking any medication that is excluded.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Lakes, PhD, Principal Investigator — UC Irvine
Locations (1):
- University of California, Irvine Child Development Center, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wigal SB, Maltas S, Crinella F, Stehli A, Steinhoff K, Lakes K, Schuck S. Reading performance as a function of treatment with lisdexamfetamine dimesylate in elementary school children diagnosed with ADHD. J Atten Disord. 2012 Jan;16(1):23-33. doi: 10.1177/1087054710378008. Epub 2010 Oct 26. PMID 20978273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through flyers and other advertising and were seen in a researach clinic setting. Subjects were recruited from july 2008 until May 2009. A primary diagnosis of ADHD was confirmed.
  All subjects were also given a K-BIT intelligence test and had to achieve a score of at least 80 to be enrolled.
Pre-assignment Details: All subjects who met study criteria for ADHD and intellectual ability who were also healthy and had no other co-morbid diagnosis except possible ODD were enrolled in the study. Any subjects taking stimulant medication before the trial did a 2-day washout before baseline. 42 subjects consented, 5 didn't meet criteria, 9 withdrew consent.
Groups:
- ADHD With Vyvanse Treatment: All enrolled subjects will be titrated to an effective dose of vyvanse. Reading abilities were tested in a modified lab school day.
Period: Vyvanse Dose Titration
Arm/Group | ADHD With Vyvanse Treatment
Started | 28
Completed | 26
Not Completed | 2
Period: Modified Lab School, Reading Evaluation
Arm/Group | ADHD With Vyvanse Treatment
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects who met study criteria for ADHD as a primary diagnosis and no other major psychiatric diagnosis and had an IQ score at 80 or above and continued to be willing to participate in Vyvanse treatment phase. All subjects received their first reading tests at baseline visit.
Arm/Group | ADHD With Vyvanse Treatment
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Gray Oral Reading Rest, Fourth Edition (GORT-4)
Description: The GORT-4 evaluates oral reading rate, accuracy and comprehension. Both Forms A and B were used.Half of the subjects randomly were tested on From A at baseline and the other half were tested with Form B.
  The GORT-4 is a standardized measure/test. Scores provided are standard scores, which range from 1 to 20, with a Mean of 10 and Standard Deviation of 3. A higher score means better reading performance. There was no total score used or calculated in this study.
Time Frame: baseline and final day (lab school Assessments)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD With Vyvanse Treatment
Number analyzed (Participants) | 26
units on a scale | 8.27 (1.84)

ADVERSE EVENTS:
Time Frame: 12 weeks from initial screening through 30 days of follow-up.
Description: adverse event data were collected in weekly visits based on spontaneous parent report until final study data. Any ongoing adverse events were again assessed at the 30 day follow-up call.
Arm/Group | ADHD With Vyvanse Treatment
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

LIMITATIONS AND CAVEATS:
This is a small sample of well characterized children with ADHD who were only treated for 1 month.

In addition, we did not select for children with reading disability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No